CLINICAL TRIAL: NCT00416026
Title: Translating Research: Patient Decision Support/Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01HS010531 (AHRQ)
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Quality improvement; Patient-centered care; Acute coronary syndrome; Telephone counseling
MeSH Terms: conditions — Acute Coronary Syndrome

INTERVENTIONS:
Behavioral: Educational/Counseling/Training

SUMMARY:
The purpose of the study was to test a telephone counseling intervention for patients after leaving the hospital for a heart attack to use medication, exercise, healthy eating and smoking cessation to prevent further heart attacks.

DETAILED DESCRIPTION:
BACKGROUND: Efficacy of brief individual telephone coaching for secondary prevention behavior has been shown. However, the independent contribution of personal counseling to system-level intervention is untested. We tested a multiple-risk factor brief counseling intervention in acute coronary syndrome (ACS) following hospital-based quality improvement (QI) program.

METHODS: Patient-level randomized trial of hospital quality improvement (QI-only) versus quality improvement plus brief telephone coaching in the first three months post-hospitalization (QI-plus) for patients hospitalized for ACS. Data collection: medical record review, state vital records, and post-hospital surveys (baseline, 3 and 8 months post hospitalization). Main outcomes: secondary prevention behaviors, physical functioning, and quality of life.

RESULTS: QI-plus patients reported statistically significant independent improvements in physical activity (OR = 1.62; p = .01) during the intervention, and were more likely to participate in formal cardiac rehabilitation (OR = 2.51; p = .02). Smoking cessation was not statistically different (OR = 1.31; p = .68); functional status and quality of life were not different at 8 months. Medication use was high in QI and QI-plus groups, and improved over prior cohorts in the same hospitals.

CONCLUSION: QI improved physician and patient adherence to guidelines and improved medical therapy in-hospital continued in the outpatient setting. Brief telephone coaching was modestly effective in accomplishing short-term, but not long-term life-style behavior change. Patient life-style behavior change appears to require sustained intervention. QI-based improvement in medication use improves survival and appears to be the most efficient route to improved outcomes for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. age of 21 years or older,
2. a documented serum Troponin I level of greater than, or equal to the upper limits of normal in each hospital, and
3. a working diagnosis of ACS in the medical record.

Exclusion Criteria:

1. inability to speak English or to complete the enrollment interview, and
2. discharge to a non-home setting.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304
Dates: Start 2002-01; Study Completion 2004-10

PRIMARY OUTCOMES:
Secondary prevention behaviors (smoking, exercise)
Physical functioning (Activity Status Index)
Quality of life (Euroqol EQ5D)

SECONDARY OUTCOMES:
Medication use

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Holmes-Rovner, PhD, Principal Investigator — Michigan State University
Locations (5):
- United States (5):
  - Genesys Health System, Flint, Michigan
  - Hurley Hospital, Flint, Michigan
  - McLaren Health Systems, Flint, Michigan
  - Covenant Health System, Saginaw, Michigan
  - St. Mary's Hospital, Saginaw, Michigan

REFERENCES:
- [Result] Yang Z, Olomu A, Corser W, Rovner DR, Holmes-Rovner M. Outpatient medication use and health outcomes in post-acute coronary syndrome patients. Am J Manag Care. 2006 Oct;12(10):581-7. PMID 17026412
- [Result] Stommel M, Olomu A, Holmes-Rovner M, Corser W, Gardiner JC. Changes in practice patterns affecting in-hospital and post-discharge survival among ACS patients. BMC Health Serv Res. 2006 Oct 24;6:140. doi: 10.1186/1472-6963-6-140. PMID 17062154
- [Result] Dunn SL, Corser W, Stommel M, Holmes-Rovner M. Hopelessness and depression in the early recovery period after hospitalization for acute coronary syndrome. J Cardiopulm Rehabil. 2006 May-Jun;26(3):152-9. doi: 10.1097/00008483-200605000-00007. PMID 16738453
- [Result] Holtrop JS, Corser W, Jones G, Brooks G, Holmes-Rovner M, Stommel M. Health behavior goals of cardiac patients after hospitalization. Am J Health Behav. 2006 Jul-Aug;30(4):387-99. doi: 10.5555/ajhb.2006.30.4.387. PMID 16787129
- [Derived] Olomu AB, Corser WD, Stommel M, Xie Y, Holmes-Rovner M. Do self-report and medical record comorbidity data predict longitudinal functional capacity and quality of life health outcomes similarly? BMC Health Serv Res. 2012 Nov 14;12:398. doi: 10.1186/1472-6963-12-398. PMID 23151237
- [Derived] Corser W, Sikorskii A, Olomu A, Stommel M, Proden C, Holmes-Rovner M. "Concordance between comorbidity data from patient self-report interviews and medical record documentation". BMC Health Serv Res. 2008 Apr 16;8:85. doi: 10.1186/1472-6963-8-85. PMID 18416841